CLINICAL TRIAL: NCT00308854
Title: PD P 506 A or Its Placebo in Combination With Red Light for Photodynamic Therapy of Mild to Moderate Actinic Keratosis
Brief Title: Photodynamic Therapy With PD P 506 A Compared With Placebo-PDT for the Treatment of AK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: photonamic GmbH & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK 03; EudraCT Number 2005-003555-13
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Actinic Keratosis
Keywords: AK; PDT
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): PD P 506 A-PDT
  Interventions: Procedure: Photodynamic Therapy
- 2 (Placebo Comparator): Placebo-PDT
  Interventions: Procedure: Photodynamic Therapy

INTERVENTIONS:
Procedure: Photodynamic Therapy

SUMMARY:
The aim of this study is to investigate whether PD P 506 A-PDT is effective in treating mild to moderate AK lesions located on the head.

DETAILED DESCRIPTION:
Actinic keratosis (AK) is a pre-cancerous skin abnormality usually caused by sun exposure. Actinic keratoses occur most commonly in fair skin, especially in the elderly. They mainly occur in sun-exposed skin areas like head and hands. It is standard of care to remove AK when diagnosed, which can be achieved by either physical ablation, chemotherapeutic agents or photodynamic therapy (PDT). A direct comparison versus placebo which is necessary for the exact quantification of the effect of PD P 506 A has not yet been performed and is subject of this study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Caucasian patients
* Diagnosis of actinic keratosis (AK) with at least three locally separated lesions located on head and/or face (hairless areas)
* Selected AK study lesions have clearly defined margins and are mild to moderate
* The distance between the study lesion borders is > 1.0 cm
* Maximum diameter of each study lesion is 1.8 cm
* Skin sun sensitivity type I to IV according to Fitzpatrick

Exclusion Criteria:

* PDT Non-responder
* Pre-treatment of the AK lesions eligible for study procedures with pharmaceuticals approved for the treatment of AK during the 4 weeks preceding PDT
* Pre-treatment of the AK lesions eligible for study procedures during the 2 weeks preceding PDT with keratolytic agents e.g. TCA, urea or salicylic acid containing formulations
* Pre-treatment with hypericin during the 2 weeks preceding PDT
* Treatment with systemic retinoids during the 3 months preceding PDT
* Treatment with cytostatics or radiation during the 3 months preceding PDT
* Female patients of childbearing potential
* Patients with clinically relevant suppression of the immune system
* Diagnosis of Porphyria
* Skin diseases that might interfere with response evaluation of study PDT
* Skin sun sensitivity type V or VI according to Fitzpatrick
* Known intolerance to one or more of the ingredients of the study medication
* Dementia or psychic condition that might interfere with the ability to understand the study and thus give a written informed consent
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding inclusion
* Suspected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Complete clinical clearance rate (CCR) of treated actinic keratosis lesions 12 weeks after PDT | 12 weeks

SECONDARY OUTCOMES:
CCR on patient basis 12 weeks, 6, 9 and 12 months after PDT | 12 months
CCR of treated actinic keratosis lesions 6, 9 and 12 months after PDT | 12 months
Adverse events/reactions and local reactions during application of the study medication as well as during and after study therapy | 12 months
Satisfaction and independent cosmetic rating of the cleared study lesions by patient and investigator in case of successful clearance and no recurrence of the lesion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Axel Hauschild, Professor MD, Principal Investigator — Christian-Albrechts-Universität zu Kiel, Germany
Locations (7):
- Germany (7):
  - Praxis Dr. Popp Dipl.-Med. Weber, Augsburg
  - Dermatologisches Zentrum Berlin, Berlin
  - Praxisklinik Professor Dr. Uwe Reinhold, Bonn
  - Zentrum Dermatologie und Venerologie, Klinikum und Fachbereich Medizin, Frankfurt a.M.
  - SciDerm, Hamburg
  - Dermatologisches Ambulatorium Hamburg-Alstertal, Hamburg
  - Gemeinschaftspraxis Dres. Scholz/Sebastian/Schilling, Mahlow